CLINICAL TRIAL: NCT03727464
Title: Memory Priming for Abstract and Concrete Words in General BIS Guided Propofol vs. Sevoflurane Anesthesia
Brief Title: Memory Priming in General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Eleonora Orena, PhD, Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AR-INNCB-PRIMING-2012
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Unconscious (Psychology)
Keywords: Memory priming; Anesthesia; Language processing; Abstract and Concrete words; Neural correlates
MeSH Terms: conditions — Unconsciousness | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Propofol Abstract Priming (Experimental): Patients undergoing propofol general anesthesia and stimulation with a list of abstract words
  Interventions: Behavioral: Abstract priming; Drug: Propofol
- Propofol Concrete Priming (Experimental): Patients undergoing propofol general anesthesia and stimulation with a list of concrete words
  Interventions: Behavioral: Concrete priming; Drug: Propofol
- Propofol Controls (Active Comparator): Patients undergoing propofol anesthesia without any intraoperative priming
  Interventions: Behavioral: Controls; Drug: Propofol
- Sevoflurane Abstract Priming (Experimental): Patients undergoing sevoflurane general anesthesia and stimulation with a list of abstract words
  Interventions: Behavioral: Abstract priming; Drug: Sevoflurane
- Sevoflurane Concrete Priming (Experimental): Patients undergoing sevoflurane general anesthesia and stimulation with a list of concrete words
  Interventions: Behavioral: Concrete priming; Drug: Sevoflurane
- Sevoflurane Controls (Active Comparator): Patients undergoing sevoflurane general anesthesia without any intraoperative priming
  Interventions: Behavioral: Controls; Drug: Sevoflurane

INTERVENTIONS:
Behavioral: Abstract priming — Patients were primed with a list of abstract during their general anesthesia
  Arms: Propofol Abstract Priming; Sevoflurane Abstract Priming
Behavioral: Concrete priming — Patients were primed with a list of concrete during their general anesthesia
  Arms: Propofol Concrete Priming; Sevoflurane Concrete Priming
Behavioral: Controls — Patients did not receive any specific stimulation with words during their general anesthesia
  Arms: Propofol Controls; Sevoflurane Controls
Drug: Propofol — Propofol general anesthesia
  Arms: Propofol Abstract Priming; Propofol Concrete Priming; Propofol Controls
Drug: Sevoflurane — Sevoflurane general anesthesia
  Arms: Sevoflurane Abstract Priming; Sevoflurane Concrete Priming; Sevoflurane Controls

SUMMARY:
Memory priming under general anesthesia is a phenomenon of incredible interest in the study of consciousness and unconscious cognitive processing, and for clinical practice.

However results from anesthesiological literature are divergent and methodologies vary.

To overcome these limits, the present study aims at better defining the phenomenon of memory priming under general anesthesia, manipulating as experimental variables both the anesthetic drug used and the stimuli primed.

DETAILED DESCRIPTION:
Some patients may develop serious psychological sequelae after surgical intervention under general anesthesia due to implicit memory formation of intraoperative events.

A number of studies in the field of anesthesiology have tried to better define the phenomenon of implicit memory in general anesthesia, with conflicting results. While some studies demonstrated the existence of unconscious memory formation also under adequate general anesthesia (BIS ranging 40-60), others state that implicit memory formation is possible only during light sedation, and that, therefore, traumatic disorders due to unconscious intraoperative memories are imputable to inadequate anesthesiological intraoperative management. The methodologies used by these studies, however, are very heterogeneous, and often inaccurate from a cognitive point of view. Data from cognitive neuroscience, in fact, demonstrate that different linguistic material, e.g. abstract and concrete words, are processed and retrieved via different networks in the brain. Then, since different anesthetics are known to target different areas of the brain, it is assumable that implicit memory formation is influenced both by the specific drug used and by the type of stimuli primed.

Therefore in this experiment, the investigators aim at testing implicit memory for different word category, abstract vs. concrete words, in patients undergoing either propofol or sevoflurane general anesthesia. Also, a very strict methodology was used both for the construction of the stimuli and the stimulation and testing procedure, in order to maximize the priming effect and exclude the risk of false positive results. The investigators hypothesize that, considering the existing data on propofol and sevoflurane effects on the brain, and the known neural correlates for abstract and concrete word processing, the priming effect would be different for abstract and concrete words between patients under propofol or sevoflurane anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing general anesthesia for back surgery
* American Society of Anesthesiology (ASA) physical status classification I or II
* Italian native speaker
* right handed (assessed with the Edinburgh Handedness Inventory)
* not to suffer from memory deficits, hearing impairment or any other medical/psychiatric condition that could affect the memory performance or hearing

Exclusion Criteria:

* to develop a postoperative cognitive dysfunction or delirium or any other medical complication that could prevent the memory testing or that could affect memory performance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-15 (Actual)

PRIMARY OUTCOMES:
Implicit score | 24 hours
  Implicit memory is tested through a word stem completion test, in which the participant has to complete a three-letter stem with the first word that comes to mind. The completion test comprises both target stems (stems of word primed intra-operatively) and foils. The number of correct completions of target stems and foils is recorded as target and non target hits. The implicit score is then calculated as (target hits - nontarget hits)/total target stimuli. The score can therefore range (absolute values) from -1 to +1, where a positive score indicates memory priming.

SECONDARY OUTCOMES:
Explicit recall of intraoperative words | before discharge from the Recovery Room and at 24 hours
  The number of intraoperative primed words that the patient is able to recall without any cue
Explicit recall of intraoperative events | before discharge from the Recovery Room and at 24 hours
  The explicit recall of intraoperative events assessed with the Brice Interview
Target hits | 24 hours
  The number of correct stem completions (hits) with target words (i.e. words heard intraoperatively)
Nontarget hits | 24 hours
  The number of correct stem completions (hits) with nontarget words (i.e. words not heard intraoperatively)

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora F Orena, PhD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orena EF, Landucci F, Ayadi R, Caldiroli D, Papagno C. Propofol and sevoflurane affect intra-operative memory formation of words differently: A prospective cohort study. Eur J Anaesthesiol. 2021 Mar 1;38(Suppl 1):S50-S57. doi: 10.1097/EJA.0000000000001417. PMID 33399379